CLINICAL TRIAL: NCT04337879
Title: A Phase Ib Study to Evaluate the Efficacy and Safety of AL2846 Capsule Combined With Chemotherapy (mFOLFOX6 or FOLFIRI)Versus Placebo Combined With Chemotherapy in Subjects With Advanced Colorectal Cancer
Brief Title: A Study of AL2846 Capsule Combined With Standard Chemotherapy Regimen in Subjects With Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL2846-I-0004
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-01

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL2846 + mFOLFOX6 (Experimental): AL2846 capsule administered orally,once daily in 28-day cycle; oxaliplatin 85mg/ ㎡ administered intravenously (IV) on day 1, day 15 in 28-day cycle；calcium folate 400mg/ ㎡ IV on day 1, day 15 in 28-day cycle；5-fu 2800mg/ ㎡ IV on day 1, 2, 15, 16 in 28-day cycle.
  Interventions: Drug: AL2846; Drug: Calcium folate; Drug: 5-FU; Drug: Oxaliplatin
- AL2846 + FOLFIRI (Experimental): AL2846 capsule administered orally,once daily in 28-day cycle; irinotecan 180mg/㎡ administered intravenously (IV) on day 1,15 in 28-day cycle; calcium folate 400mg/ ㎡ IV on day 1,15 in 28-day cycle; 5-fu 2800mg/ ㎡ IV on day 1, 2, 15, 16 days in 28-day cycle.
  Interventions: Drug: AL2846; Drug: Calcium folate; Drug: 5-FU; Drug: Irinotecan

INTERVENTIONS:
Drug: AL2846 — AL2846 is a multi-target receptor tyrosine kinase inhibitor, which has obvious selectivity for c-met.
Drug: Calcium folate — Calcium folate 400mg/ ㎡ IV on day 1,15 in 28-day cycle
Drug: 5-FU — 5-FU 2800mg/ ㎡ IV on day 1, 2, 15, 16 days in 28-day cycle.
Drug: Oxaliplatin — Oxaliplatin 85mg/ ㎡ administered intravenously (IV) on day 1, day 15 in 28-day cycle.
  Arms: AL2846 + mFOLFOX6
Drug: Irinotecan — Irinotecan 180mg/㎡ administered intravenously (IV) on day 1,15 in 28-day cycle.
  Arms: AL2846 + FOLFIRI

SUMMARY:
This is a study to explore the safety, tolerance and efficacy of AL2846 capsules combined with mFOLFOLX6 or FOLFIRI standard chemotherapy regimen in subjects with advanced metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

-1. Histologically confirmed advanced metastatic colorectal cancer. 2. Has received only first-line standard chemotherapy regimen for metastatic disease, and which was failed.

3. At least one measurable lesion. 4. Has received systemic chemotherapy, palliative radiotherapy or other anti-tumor therapy before first dose at least 4 weeks.

5.18 and 75 years old; Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.

6. Adequate laboratory indicators. 7. No pregnant or breastfeeding women, and a negative pregnancy test. 8. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Diagnosed and/or treated additional malignancy within 5 years with the exception of basal cell carcinoma of the skin and carcinoma in situ of the cervix.

  2. Has received radiotherapy, chemotherapy and surgery before and less than 4 weeks from the first administration and less than 5 half-lives of oral targeted drugs after the completion of treatment.

  3. Has multiple factors that affect oral medications. 4. Has gastroduodenal ulcer, ulcerative colitis, intestinal obstruction and other gastrointestinal diseases or other conditions judged by the investigator that may cause gastrointestinal bleeding or perforation.

  5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.

  6. Has arterial or deep vein thrombosis events in 6 months. 7. Hypersensitivity to AL2846 or its excipient. 8. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear.

  9. Has symptomatic brain metastases, spinal cord compression, and cancerous meningitis within 8 weeks,or brain or pia mater disease confirmed by CT or MRI examination before the first dose.

  10.Has adverse events caused by previous therapy that did not recover to ≤ grade 1, with the exception of alopecia or ≥ grade 2 neurotoxicity caused by Oxaliplatin.

  11. Subjects plan to receive FOLFIRI chemotherapy regimen with uridine diphosphate glucuronyltransferase homozygous variant or double hybrid variant.

  12. Has drug abuse history that unable to abstain from or mental disorders. 13. Has any serious and/or uncontrolled disease. 14. Has received allogeneic organ transplants, hematopoietic stem cell transplants or bone marrow transplants.

  15. Has participated in other clinical trials within 4 weeks before the first dose.

  16. According to the investigators' judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 12 month
  PFS defined as the time from the first dose until the first documented progressive disease (PD) or death from any cause, based on investigator.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 12 month
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | up to 12 month
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of response (DOR) | up to 12 month
  The time when the participants first achieved complete or partial remission to disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shengyang, Liaoning, China